CLINICAL TRIAL: NCT04668456
Title: The Effect of Subtenon and Intravenous Dexmedetomidine on Patients Undergoing Cataract Surgery: A Comparative Randomized Controlled Double Blind Study
Brief Title: Subtenon and Intravenous Dexmedetomidine Effect on Patients Undergoing Cataract Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, ashraf magdy eskandr, assistant professor of anesthesia, icu, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8/8/2020 ANET4
Record Dates: First submitted 2020-12-02; First posted 2020-12-16 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Acute Postoperative Pain
Keywords: subtenon; dexmedetomidine; cataract surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: 75 Patients were assigned into three equal groups, all patients received 2.5 ml of local anesthetic mixture through subtenon block and IV infusion of drugs as follows: Group C (control group): received subtenon LA mixture of bupivacaine 0.5% (1 ml) + lidocaine 2% (1 ml)+ saline 0.9% (0.5 ml) and IV infusion of saline 0.9% over 10 min. before subtenon block.
  Group SD ( subtenon dexmedetomidine): received subtenon LA mixture of bupivacaine 0.5% (1 ml) + lidocaine 2% (1 ml)+ 0.5 μg/kg dexmedetomidine (0.5 ml) and IV infusion of saline 0.9% over 10 min. before subtenon block.
  Group ID (iv dexmedetomidine): received received subtenon LA mixture of bupivacaine 0.5% (1 ml) + lidocaine 2% (1 ml)+ saline 0.9% (0.5 ml) and IV infusion of 0.5 μg/kg dexmedetomidine over 10 min. before subtenon block.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group C (control group) (Placebo Comparator): Group C (control group): received subtenon LA mixture of bupivacaine 0.5% (1 ml) + lidocaine 2% (1 ml)+ saline 0.9% (0.5 ml) and IV infusion of saline 0.9% over 10 min. before subtenon block.
  Interventions: Drug: lidocaine 2%; Drug: bupivacine 0.5%; Drug: Normal saline
- Group SD (subtenon dexmedetomiine) (Active Comparator): Group SD ( subtenon dexmedetomidine): received subtenon LA mixture of bupivacaine 0.5% (1 ml) + lidocaine 2% (1 ml)+ 0.5 μg/kg dexmedetomidine (0.5 ml) and IV infusion of saline 0.9% over 10 min. before subtenon block.
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine 2%; Drug: bupivacine 0.5%; Drug: Normal saline
- Group ID (iv dexmedetomidine) (Active Comparator): Group ID (iv dexmedetomidine): received received subtenon LA mixture of bupivacaine 0.5% (1 ml) + lidocaine 2% (1 ml)+ saline 0.9% (0.5 ml) and IV infusion of 0.5 μg/kg dexmedetomidine over 10 min. before subtenon block.
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine 2%; Drug: bupivacine 0.5%

INTERVENTIONS:
Drug: Dexmedetomidine — the drug administered either subtenon ot iv
  Arms: Group ID (iv dexmedetomidine); Group SD (subtenon dexmedetomiine)
Drug: lidocaine 2% — subtenon injection
Drug: bupivacine 0.5% — subtenon injection
Drug: Normal saline — either subtenon or iv
  Arms: Group C (control group); Group SD (subtenon dexmedetomiine)

SUMMARY:
The study designed to compare the effects and the safety of adding dexmedetomidine to local anesthetics and its intravenous administration in subtenon block in patients undergoing cataract surgery.

DETAILED DESCRIPTION:
Ophthalmological surgery can be performed under topical, regional or general anesthesia. Recently, the majority of ocular surgeries performed by regional rather than general anesthesia, because of the regional anesthesia is more economic, easy to perform, and the risk involved is less. Orbital regional anesthesia can be done using a retrobulbar (intra-conal) block, peribulbar (extra-conal) block or sub-Tenon's block.

The STBs or episcleral block was first described by Turnbull in 1884 and it was repopularized in the 1990s as a simple and safe alternative to needle-based eye blocks. The STB becomes the most widely practiced regional technique for cataract surgery, because it produces satisfactory anesthesia for most intraocular procedures, and avoids the inherent risks of needle-based blocks, such as globe perforation and optic nerve injury.

Dexmedetomidine is a selective α-2 receptor agonist that produces sedation and analgesia without causing respiratory depression. It also allows patients to respond to verbal commands during the sedation; easy conversion from sleeping to awakening is possible. Therefore, dexmedetomidine has been used as sedative in various clinical fields in intensive care unit and surgery and an adjuvant to local anesthetics.

Many studies were done to evaluate its effect as sedative or anlgesic when administered either intravenously or when added to local anesthesia in ophthalmic block. But no one, till now comparing its effect when used as adjuvant to local anesthetics or administered intravenously in subtenon block.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-III
* Aged 18-70 years
* Both sex
* Scheduled for elective phacoemulsification cataract surgery

Exclusion Criteria:

* Coagulation abnormalities
* Impaired mental status
* Refusal of the patient
* Uncontrolled glaucoma
* Recent surgical procedure on the same eye

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-03-14 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
duration of sensory block | 24 hours
  time from injection of local anesthetic mixture to complete recovery from pain sensation or the first need of rescue analgesia

SECONDARY OUTCOMES:
duration of motor block | 24 hours
  time from injection of local anesthetic to complete recovery of motor function in all ocular muscles.

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - Ashraf magdy Eskandr, Shibīn al Kawm, Monufia Governorate
  - Osama A Elmorsy, Shibīn al Kawm, Monufia Governorate
  - Sadik A Sadik, Shibīn al Kawm, Monufia Governorate

IPD SHARING:
Plan to Share IPD: No